CLINICAL TRIAL: NCT05433415
Title: Black Girls Move: A Daughter/Mother Intervention to Prevent Obesity by Increasing Physical Activity and Improving Dietary Intake Among Black Adolescent Daughters
Brief Title: Black Girls Move Physical Activity and Improving Dietary Intake Among Black Adolescent Daughters
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Illinois at Chicago (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK132698 (NIH); R01DK132698 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Adolescent Obesity; Diabetes Mellitus
Keywords: dyad; mothers; daughters; physical activity; nutrition; racism
MeSH Terms: conditions — Pediatric Obesity; Diabetes Mellitus; Motor Activity; Racism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black Girls Move (BGM) Treatment Condition (Experimental): BGM is guided by the Anti-Racist Public Health Critical Race Praxis with adaptive mechanisms to support Black adolescent females as they navigate a racist society. The BGM treatment condition will include mothers as active participants in all components of the weekly, 12-session intervention to test the impact of actively leveraging the daughter/mother relationship . Participants in our prior research endorsed the importance of daughters and mothers actively engaging in group meetings together on weekends. Participants set PA and diet goals and self-monitor goal attainment. Dyads participate in structured activities designed to facilitate communication, problem solving, role assignment, and relationship quality. Dyads use a variety of videos, role play, discussion, and activities to achieve session outcomes. The sessions are led by trained facilitators who follow a standardized facilitator manual.
  Interventions: Behavioral: Black Girls Move
- Daughters-Only Comparison Condition (DOCC) (Active Comparator): The DOCC runs parallel to the BGM intervention and includes daughters-only group meetings. The DOCC incorporates all components of BGM except Family Systems Theory strategies. Daughters in DOCC will receive PA and diet behavior content based on Anti-Racist Public Health Critical Race Praxis and Social Cognitive Theory with daughter-only group activities. DOCC facilitators will lead group meetings and discussions. All DOCC daughters will self-monitor their progress towards PA goals using Fitbit® and progress towards diet goals using Start Simple with My Plate®.
  Interventions: Behavioral: Black Girls Move

INTERVENTIONS:
Behavioral: Black Girls Move — Goal setting and monitoring. All BGM daughters will self-monitor their progress towards PA goals using a PA device, Fitbit®. Additionally, BGM daughters will self-monitor their progress towards diet goals using a mobile application, Start Simple with My Plate®. Further, all BGM mothers will use Fitbit® and Start Simple with My Plate® for self monitoring, however, mothers' data will not be analyzed for this study. Since the daughter/ mother relationship is critical to achieving behavioral change, BGM mothers will utilize Fitbit® and Start Simple with My Plate® as a mechanism to communicate, problem solve and support daughters' behavioral goals.BGM is situated within the contexts of environmental, cultural, interpersonal, and developmental factors impacted by structural racism. Intentionally engaging mothers and daughters in an asset based program provides a framework for mothers to model responses to structural racism i.e. racial socialization.

SUMMARY:
Black Girls Move is a school-linked daughter/mother physical activity and dietary behavior program, with 9th and 10th grade students. This program is designed to prevent obesity in Black adolescent females and thus aligns with the NIH mission to enhance health, lengthen life, and reduce illness and disability. This project is relevant to public health because it holds the potential to reduce population health disparities impacted by structural racism.

DETAILED DESCRIPTION:
Black female adolescents are at increased risk for obesity-related morbidity and mortality as adults compared to non-Hispanic White female adolescents. Interventions to prevent obesity in Black female adolescents that leverage the relationship of the daughter/mother dyad have received limited attention. Studies that do include mothers tend to use theoretical frameworks that do not explicitly build on this important family relationship and have not included mothers' active participation. Additionally, these studies do not include girls over the age of 12. In response, the investigators developed Black Girls Move, a school-based obesity prevention intervention that addresses these limitations in the extant literature. The investigators conducted focus groups with daughter/mother dyads to identify practical, cultural, and age-appropriate strategies for improving physical activity (PA) and dietary behaviors in Black adolescent daughters (grades 9-10, ages 14-17). Black Girls Move consists of 12 weekly group sessions of daughter/mother dyads in which participants set individualized PA and dietary goals. Black Girls Move incorporates content and processes derived from asset-based anti-racist Public Health Critical Race Praxis, Family Systems Theory, and Social Cognitive Theory. Specific aims are to determine the efficacy of Black Girls Move compared to daughters-only comparison condition on change in PA and dietary intake, and the impact of Black Girls Move compared to daughters-only on theoretical mechanisms of change (racial identity, daughter/mother relationship, social cognitions) assessed by self-report measures.

The design is a 12-week pre-test/post-test, randomized controlled trial. The investigators will recruit 24 daughter/mother dyads at each of 8 schools for a total sample size of 192 daughter/mother dyads (total 384 participants). Within school, each dyad will be randomized to either Black Girls Move or daughters-only comparison condition (12 per condition). All daughters and all mothers (Black Girls Move daughter/mother dyads and daughters-only comparison condition daughter/mother dyads) complete assessments (e.g., PA, diet, family measures) at baseline, post-intervention, and 3-months post-intervention. The investigators recognize that there are potential validity threats associated with within school student randomization. The investigators will collect data to assess the degree to which these potential threats are pertinent. The long-term goal of this research is to decrease disparities in obesity and associated comorbidities in Black women. The findings may inform future large scale R01 studies of BGM in Black daughter/mother dyads

ELIGIBILITY:
Inclusion Criteria for daughters are:

* English speaking;
* Black;
* grade 9 or 10;
* daily access to the internet outside of school and/or work through an iOS or android smart phone, tablet, or personal computer;
* either high-normal weight (between ≥50th and <85th percentile for age and gender) or overweight (between ≥85th and <95th percentile for age and gender) as the purpose of this study is weight maintenance and obesity prevention in at-risk daughters rather than obesity treatment; 98 and
* have either a poor diet, (defined as consuming <1 vegetable or <1 fruit per day) 99 or inadequate PA (defined as < 60 minutes per day, 7 days per week). 99,100

Inclusion criteria for mothers are:

* English-speaking;
* Black;
* co-residing biological mother or mother-figure and legal guardian of the participating daughter;
* the person primarily responsible for meals in the household; and
* access to the internet through an iOS or android smart phone, tablet or personal computer. In a longitudinal study of 480 adults, 84% of adults with obesity were adolescents with high normal weight status (≥50th and <85th percentile). National data on cell phone ownership show that 81% of Black students and 68% of Black parents own a smart phone

Exclusion Criteria:

The exclusion criteria for both daughters and mothers includes:

* having conditions/procedures that prevent the oral consumption of foods (e.g., gastric feeding tubes);
* presence of physical limitations that would preclude participation in the PA activity components of the intervention;
* altered dietary intake (e.g., pregnancy, eating or metabolic disorders except for type 1 or type 2 diabetes); and
* at baseline physical assessment, participants screened for uncontrolled blood pressure (systolic > 130, diastolic >80 for daughters; and systolic >160, diastolic >100 for mothers) will be eligible only with a healthcare provider release.
* participants with diagnosed type 1 or 2 diabetes will be eligible for participation only with a healthcare provider release.
* mothers will be screened for cardiovascular disease and musculoskeletal risk factors with the 7-item Physical Activity Readiness Questionnaire. Mothers that answer 'yes' to any item on the Physical Activity Readiness Questionnaire will be eligible only with a healthcare provider release. Daughters or mothers who are asked to provide healthcare provider release will be referred to the Chicago Department of Public Health if they do not have a primary care provider. To be eligible to participate in either condition, both the daughter and her mother must be willing and eligible to participate in the study.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Actigraph GT3X Device at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  Objective measure of daughter and mother daily steps and activity counts. PA levels operationalized as moderate (1500-2600 counts/30 secs) or vigorous (>2600 count/30 secs). Device worn for one week during waking hours
Change from Block Kids 2004 Food Frequency Questionnaire (BKFFQ) at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 72-item self-report measure of daughter dietary behavior over the past week. Participants indicate frequency of consumption of food/beverages on a 6-point scale (none to every day).

SECONDARY OUTCOMES:
Change from 3-Day Physical Activity Recall at 12 and 24 weeks moderate/vigorous physical activity per week | Baseline, 12 weeks, and 24 weeks
  A 59-item self-report measure of daughter physical activity. Participants recall 59 physical activity activities in the past 3 days. Each day divided into 34, 30-minute blocks from 7 am to midnight. Activities rated as light, moderate, hard, or very hard.
Change from The Multidimensional Model of Black Identity - Short Form at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 27-item self-report measure of daughter and mother racial identity.
Change from Child Health Behavior Knowledge Scale at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 9-item self-report measure of daughter and mother physical activity knowledge related to cardiovascular benefits of exercise.
Change from Diet and Health Knowledge Survey at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 42-item self-report measure of daughter and mother diet knowledge.
Change from Physical Activity and Nutrition Self-Efficacy Scale at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  An 11-item self-report measure of daughter self-efficacy for physical activity (3 items) and nutrition (8 items) behaviors.
Change from Social Support for Physical Activity at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  An 11-item self-report measure of daughter social support for physical activity.
Change from Social Support Scale at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 5-item self-report measure for daughter and mother social support for healthy eating.
Change from Family Assessment Device (FAD) at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 53-item self-report measure of daughter and mother perceptions of family systems.
Change fron Quality of Mother Interaction at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 14-item self-report measure of daughter perceptions of quality of communication with mother

OTHER OUTCOMES:
Two-Item Hunger VitalSignTM | Baseline
  A 2-item self-report questionnaire evaluating daughter and mother food insecurity in the past 12 months.
Change from International Physical Activity Questionnaire at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 27-item self-report measure of mother physical activity. Activities pertain to job (7), transportation (6), household (6), recreation (6), and sitting (2). Participants indicate frequency (days), duration (hours/minutes), and intensity (moderate to vigorous) over past 7days.
Change from 2014 Block Food Frequency Questionnaire at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 127-item self-report measure of mother dietary behavior. Items similar to BKFFQ with additional items to adjust for fat, protein, carbohydrate, sugar, and whole grain content
Change from Self-Efficacy for Walking Scale at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 12-item self-report measure of mother self-efficacy for walking.
Change from Weight Efficacy Lifestyle Questionnaire at 12 and 24 weeks | Baseline, 12 weeks, and 24 weeks
  A 20-item self-report measure of mother dietary self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Reed, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reed M, Wilbur J, Tangney CC, Miller AM, Schoeny ME, Webber-Ritchey KJ. Development and Feasibility of an Obesity Prevention Intervention for Black Adolescent Daughters and Their Mothers. J Healthy Eat Act Living. 2021 Apr 1;1(2):94-107. eCollection 2021. PMID 37789909
- [Background] Reed M, Julion W, McNaughton D, Wilbur J. Preferred intervention strategies to improve dietary and physical activity behaviors among African-American mothers and daughters. Public Health Nurs. 2017 Sep;34(5):461-471. doi: 10.1111/phn.12339. Epub 2017 Jun 22. PMID 28639382
- [Background] Reed M, Wilbur J, Schoeny M. Parent and African American Daughter Obesity Prevention Interventions: An Integrative Review. J Health Care Poor Underserved. 2015 Aug;26(3):737-60. doi: 10.1353/hpu.2015.0103. PMID 26320909

DOCUMENTS (1):
  • Informed Consent Form (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/15/NCT05433415/ICF_001.pdf